CLINICAL TRIAL: NCT05322148
Title: The CLEAN Study: Cyclosporine 0.1% / Loteprednol 0.2% Effect on Anterior Segment Normalization-A Prospective Cohort Study of Combination Therapy in the Treatment of Dry Eye
Brief Title: Cyclosporine 0.1% / Loteprednol 0.2% Effect on Anterior Segment Normalization
Acronym: CLEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010 CLEAN Klarity CL
Record Dates: First submitted 2022-02-17; First posted 2022-04-11 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Loteprednol Etabonate

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, randomized controlled, open label study of the efficacy of cyclosporine 0.1% / loteprednol 0.2% in improving higher order aberrations, and TBUT in patients with dry eye. Patients will be randomized to receive treatment with either cyclosporine 0.1% / loteprednol 0.2% BID for 4 weeks or cyclosporine 0.05% BID for 4 weeks and will be evaluated at baseline (before treatment), 14 days, and 28 days of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cyclosporine 0.1% / loteprednol 0.2% group (Active Comparator): 60 total patients will be randomized in a 2 to 1 proportion with 40 in the cyclosporine 0.1% / loteprednol 0.2% group and 20 in the cyclosporine 0.05% group. All patients will undergo treatment in both eyes.
  Interventions: Drug: Klarity CL, Cylcosporine 0.1%/Loteprednol Etabonate 0.2% Preservative Free
- cyclosporine 0.05% group (Active Comparator): 60 total patients will be randomized in a 2 to 1 proportion with 40 in the cyclosporine 0.1% / loteprednol 0.2% group and 20 in the cyclosporine 0.05% group. All patients will undergo treatment in both eyes.
  Interventions: Drug: Klarity CL, Cylcosporine 0.1%/Loteprednol Etabonate 0.2% Preservative Free

INTERVENTIONS:
Drug: Klarity CL, Cylcosporine 0.1%/Loteprednol Etabonate 0.2% Preservative Free — A number of studies have shown the benefit of both cyclosporine and steroids in managing dry eye. However, existing formulations of these products are challenged by either limited tolerability, a high out-of-pocket cost or both. Combination therapy with these agents in an advanced, more tolerable formulation have the potential to improve both tolerability and cost. However, the available formulation of preservative free Klarity CL (cyclosporine 0.1% and loteprednol 0.2% in a chondroitin sulfate vehicle) has not been studied rigorously.

SUMMARY:
The CLEAN Study: Cyclosporine 0.1% / Loteprednol 0.2% Effect on Anterior Segment Normalization-A Prospective Cohort Study of Combination Therapy in the Treatment of Dry Eye

DETAILED DESCRIPTION:
Thirty million people in the US are thought to suffer from dry eye. Patients with this condition manifest with ocular surface disruption such as corneal fluorescein staining and reduced tear breakup time (TBUT). Successful treatment is a high priority for both patients and physicians, reducing symptoms and improving visual acuity and corneal higher order aberrations (HOAs), which have been closely linked with treatment satisfaction. A number of studies have shown the benefit of both cyclosporine and steroids in managing dry eye. However, existing formulations of these products are challenged by either limited tolerability, a high out-of-pocket cost or both. Combination therapy with these agents in an advanced, more tolerable formulation have the potential to improve both tolerability and cost. However, the available formulation of preservative free Klarity CL (cyclosporine 0.1% and loteprednol 0.2% in a chondroitin sulfate vehicle) has not been studied rigorously.

This study is designed to demonstrate that Klarity CL can benefit the ocular surface with high tolerability, making it a very desirable method of treating patients with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients over age 18 with the following signs:

  i. Central or inferior corneal fluorescein staining defined by the Oxford Scale ii. Reduced tear break up time (TBUT) ≤ 10 seconds.
* Able to comprehend and sign a statement of informed consent.
* Patients willing to take an electronic survey about their tolerability of either study medication.
* Willing and able to complete all required postoperative visits.

Exclusion Criteria:

* Ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgical procedure) performed within the last 3 months or at any time that in the investigator's clinical judgment if it would interfere with the outcome measures of this study.
* Clinically significant ocular trauma.
* Active ocular Herpes simplex or Herpes Zoster infection
* Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) at the discretion of the investigator.
* Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye).
* Active, systemic or local disease condition that causes clinically significant ocular surface irritation such that it could interfere with the study findings.
* Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis.
* Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
* Eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis).
* Ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
* Participation in this trial in the same patient's fellow eye
* Patients who are under age 18, pregnant or breastfeeding, or who may become pregnant during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Primary Study Measure - Corneal Higher Order Aberrations by Topography | Up to 2 months
  Change in corneal higher order aberrations after 14 days and 28 days of treatment

SECONDARY OUTCOMES:
Secondary Measure - SPEED Questionnaire to track progression of dry eye symptoms over time | Up to 2 months
  SPEED score at baseline, 14, and 28 days of treatment. Slit lamp exam at baseline, 2 weeks and 4 weeks to determine ocular hyperemia (Schulze Scale), tear breakup time (TBUT), cornea staining (Oxford scale)

OTHER OUTCOMES:
Exploratory Outcome Measure | Up to 28 days
  Tolerability score on modified COMTOL scale at 14, and 28 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — Harvard Eye Associates
Locations (3):
- United States (3):
  - Inland Eye Specialists, Hemet, California
  - Harvard Eye Associates, Laguna Hills, California
  - Cleveland Eye Clinic, Brecksville, Ohio

IPD SHARING:
Plan to Share IPD: Undecided